CLINICAL TRIAL: NCT06420856
Title: Is There a Relationship Between Protective Sole Sense, Ankle Proprioception, Ankle Mobility and Balance in Patients With Treated Lisfranc Injury?
Brief Title: Changes of Various Structures After Lisfranc Injury Compared to Healthy Individuals.
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ali Ilez, Research Assistant, Istanbul Saglik Bilimleri University
Other Study IDs: SBU-FTR-AI-02
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Lisfranc Injury
Keywords: Proprioception; Postural Balance; Foot Injuries
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lisfranc injury patients: Sense of light touch will be used with the Semmes-Weinstein Monofilament test, Proprioception evaluation will be used with the Dr.Goniometer application, Muscular strength and endurance will be evaluated with the cybex isokinetic device, Weight-Bearing Lunge test will be used to evaluate ankle mobility and Modified Star Excursion Balance Test will be used to evaluate dynamic balance.
  Patients' functional levels will be evaluated under two headings:
  1. Questionnaire-based functional evaluation: American Orthopedic Foot and Ankle Society (AOFAS) midfoot score and foot and ankle functions Rating Foot and Ankle Outcome Score (FAOS) will be used and will be evaluated.
  2. Physical performance evaluation: Heel raise test would be used
  Interventions: Other: Assessment of the musculoskeletal system and its functions
- Healthy Volunteers: Sense of light touch will be used with the Semmes-Weinstein Monofilament test, Proprioception evaluation will be used with the Dr.Goniometer application, Muscular strength and endurance will be evaluated with the cybex isokinetic device, Weight-Bearing Lunge test will be used to evaluate ankle mobility and Modified Star Excursion Balance Test will be used to evaluate dynamic balance.
  Patients' functional levels will be evaluated under two headings:
  1. Questionnaire-based functional evaluation: American Orthopedic Foot and Ankle Society (AOFAS) midfoot score and foot and ankle functions Rating Foot and Ankle Outcome Score (FAOS) will be used and will be evaluated.
  2. Physical performance evaluation: Heel raise test would be used
  Interventions: Other: Assessment of the musculoskeletal system and its functions

INTERVENTIONS:
Other: Assessment of the musculoskeletal system and its functions — Measurement of sub sole pressure sense, light touch sense, vibration sense and two-point discrimination sense. will be evaluated with. For the evaluation of proprioception, active joint position sense technique was used in plantar flexion (PF): 7°, 14° and 21°; In dorsiflexion (DF), 7° target angles will be used. An Dr. Goniometer will be used to determine target angles. To measure plantarflexion and dorsiflexion muscular strength and endurance will be used with the isokinetic system. Weight-Bearing Lunge test will be used to evaluate ankle mobility. For balance assessment, the Modified Star Excursion Balance Test will be measured using the anterior, posteromedial and posterolateral directions. American Orthopedic Foot and Ankle Society midfoot score and foot and ankle functions Rating Foot and Ankle Outcome Score , which are subjective evaluation methods, will be used to determine the functional level. A heel lift test will be performed to evaluate physical performance.

SUMMARY:
The effect of muscular strength deficits on postural control after Lisfranc injury has been explained in relation to stance duration and strength. However, the relationship between protective sole sensation and changes in ankle proprioception, balance, ankle mobility and Achilles tendon structural properties has been shown in previous studies. The aim of our study was to determine the possible changes in protective sole sensation, ankle proprioception, balance and functional capacity after Lisfranc injury and to analyse the relationship between these variables.

DETAILED DESCRIPTION:
'Lisfranc injury' refers to an injury in which one or more metatarsals are displaced. Lisfranc injury covers a wide network of injuries. It includes various types, including a low-energy sports injury or a high-energy lesion, as well as a purely connective tissue injury. 20% of Lisfranc injuries are undiagnosed or diagnosed late. Early and accurate diagnosis of injuries is a basic requirement for appropriate treatment and prevention of secondary problems that may arise in the long term . Fracture-dislocation in the tarsometatarsal junction of the foot is treated with anatomical reduction, internal fixation or primary arthrodesis. However, many individuals have poor functional outcomes . Anatomical repositioning and excellent postoperative radiographic findings may not result in high patient satisfaction. As a result, no matter what type of treatment is used after Lisfranc injury, it should be supported by a good rehabilitation protocol. As a result of our research in the literature, the investigators encountered studies that performed gait analysis, muscle strength and plantar pressure measurements after Lisfranc injury. However, no study has been encountered examining parameters such as sole sense, proprioception, and balance after injury of the foot, which is the only limb in contact with the ground. After determining these values, revising the rehabilitation protocols specifically for the evaluation parameters will reduce the morbidity rate after injury and accelerate functional recovery.

Rehabilitation protocols that emphasize the use of exercises to improve joint range of motion, muscle strength, neuromuscular coordination, and gait mechanics after foot and ankle injuries have been found to improve function . There is also evidence that the plantar flexor muscles of these patients are weakened after injury. There are also groups of patients who complain of instability when walking barefoot or on uneven ground after foot or ankle injuries. In a different study examining the dynamic plantar pressure distribution, force capacity and postural control change after Lisfranc injury, it was found that atrophy occurred after long-term immobilization in both the injured extremity and the contralateral extremity.

Altered postural control after injury was manifested by a significant decrease in unilateral stance time. Adequate rehabilitation following anatomical open reduction after Lisfranc injury is very important for clinical outcome. A detailed evaluation is required to determine adequate rehabilitation. Considering these studies, evaluating balance will be important for patients with Lisfranc injuries.In our study, the investigators aim to provide information about postural control change after injury by evaluating dynamic balance with the Modified star excursion test. In this way, the intensity of balance exercises can be adjusted while shaping the post-injury rehabilitation program. Evaluated gait analysis and functional results in patients following a designated rehabilitation program after Lisfranc injury. In this study evaluating patients with lisfranc injury treated with 3 different methods (conservative, open reduction internal fixation and primary arthrodesis), significantly reduced joint range of motion, lower walking speed and significantly lower flexion/extension of the midfoot compared to healthy subjects during the pushing phase. These changes may result from loss of muscle strength, differences in surgical methods or different rehabilitation protocols. This change during the pushing phase and the decrease in walking speed negatively affect the lives of patients functionally.

Determination of ankle mobility after injury, determination of rehabilitation effectiveness and functional evaluation will be used for the first time in our study for patients with lisfranc injury. In addition to this information, in our study, the investigators aim to evaluate functional capacity with AOFAS (American Orthopaedic Foot and Ankle Society) Midfoot Score , FAOS(Foot and Ankle Outcome Score) and heel-rise tests and be the first study in the literature to apply this test on ligamentous injury. The data obtained after the evaluation may increase the clinical use of these easy and inexpensive tests. Thus, function after Lisfranc injury can be evaluated much more easily, quickly and objectively. Lisfranc injury does not only cause deficits in muscle strength and joint range of motion. Many factors, such as long-term immobilization after injury, damage to structures rich in mechanoreceptors, or surgery, can lead to changes in both sole sensation and joint position sense.

ELIGIBILITY:
Inclusion Criteria for Lisfranc Injury Group:

* Having had a Lisfranc injury
* Having only one extremity injured
* Having received surgical treatment
* Being over 18 years old

Exclusion Criteria for Lisfranc Injury Group :

* Having a neurological problem,
* diabetes
* smoking
* untreated Lisfranc injury
* incomplete medical record
* not wanting to participate in the study
* having a neurovascular injury

Inclusion Criteria for Healthy Volunteer Group

* Being healthy
* Any foot pain, history of fractures, etc. Absence of circumstances
* Being over 18 years of age

Exclusion Criteria for Healthy Volunteer Group

* Not being healthy
* Any foot pain, history of fractures, etc.
* Not being over 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 24 people will be included in our study. It will be conducted with 12 Lisfranc injury patients and 12 healthy volunteer participants. All participants will be over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Difference in plantar sensation in people with Lisfranc injuries compared to healthy people | 2 months
  Our primary outcome is to determine the difference in plantar sensation changes in people with Lisfranc injuries after treatment compared to healthy volunteers with similar demographic characteristics. According to the monofilament test results, increasing numerical values indicate that proprioception is negatively affected.

SECONDARY OUTCOMES:
AOFAS (American Orthopaedic Foot and Ankle Society) midfoot Score | 1 months
  American Orthopaedic Foot and Ankle Society (AOFAS) Midfoot Rating System range from 0 to 100, with a healthy midfoot receiving 100 points. This score may be used to assess the intercuneiform, lateral cuneiform-cuboid, naviculocuneiform, and tarsometatarsal levels and may be useful for fractures and arthrodesis procedures.
FAOS (Foot and Ankle Outcome Score) Score | 1 months
  Foot and Ankle Outcome Score (FAOS) subscale scores range from 0 to max , with higher scores indicating better outcomes. A score of 100 on a subscale indicates no symptoms or limitations in that particular area, while a score of 0 indicates extreme symptoms and limitations.
Modified Star Excursion Test | 1 months
  For balance assessment, the Modified Star Excursion Balance Test will be measured using the anterior, posteromedial and posterolateral directions. Lower Extremity Normalization Score and Composite Score will be used for this measurement.Higher values indicate a better balance.

CONTACTS AND LOCATIONS:
Overall Officials: ALİ İLEZ, Principal Investigator — Istanbul Saglik Bilimleri University
Locations (1):
- İstanbul Tıp Fakültesi Ortopedi ve Travmatoloji Anabilimdalı, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No